CLINICAL TRIAL: NCT04523766
Title: Enhancing Pain Management and Preventing Opioid Misuse by Optimizing Mindfulness Based Interventions for Opioid-Treated Chronic Pain Patients: A Comparison of Mindful Interoceptive Mapping and Mindful Breathing
Brief Title: Comparing the Impact of Mindful Interoceptive Mapping and Mindful Breathing on Pain and Opioid Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Adam Hanley, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB_00135443
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Pain, Chronic; Opioid Use
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness of Breath (Active Comparator)
  Interventions: Behavioral: Mindfulness of Breath
- Mindful Interoceptive Mapping (Experimental)
  Interventions: Behavioral: Mindful Interoceptive Mapping

INTERVENTIONS:
Behavioral: Mindfulness of Breath — The Mindful Breathing intervention will be adapted from a validated, brief mindfulness training model. Participants will be instructed to focus on the sensations of the breath (i.e., at the tip of the nose and in the nostrils, abdomen and back) and, if a pain arises in the body, acknowledge it without judgement and return attention to the breath.
  Arms: Mindfulness of Breath
Behavioral: Mindful Interoceptive Mapping — The MIM intervention will be adapted from the core MORE meditation practice. Participants will be instructed to (1) zoom in to deconstruct pain into its constituent affectively-valenced physical sensations and precisely map each sensation's spatial location, (2) zoom out to broaden the field of attention to include previously neglected sensory elements (i.e., spaces within the body that are absent of sensation and pleasant sensations), and (3) savor any pleasant sensations or experiences occurring during the mindfulness practice.
  Arms: Mindful Interoceptive Mapping

SUMMARY:
This is a single site, two-arm, parallel group randomized clinical trial comparing the effect of two mindfulness-based interventions (Mindful Interoceptive Mapping vs. Mindfulness of the Breath) on opioid-treated chronic pain patients' pleasant/unpleasant sensation reports and opioid use.

ELIGIBILITY:
Inclusion Criteria:

* (1) men/women ≥18 years of age,
* (2) current chronic low back pain condition determined by physician assessment (e.g., ICD-10 codes M54.5, M54.4, M54.3),
* (3) reporting pain ≥3 on 0-10 scale with opioid medication, and
* (4) long-term opioid pharmacotherapy (>3 months of use).

Exclusion Criteria:

* (1) formal mindfulness training (e.g., MBSR/MBRP),
* (2) current cancer diagnosis,
* (3) psychosis, suicidality, and moderate/severe substance use disorder in the past year as assessed with the MINI, and
* (4) unstable illness, as judged by a physician, that may interfere with treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Immediate Change in Pleasant Sensation Ratios | Immediately before and immediately after the final mindfulness training session, approximately 30 minutes
  The Multidimensional Assessment of Pleasant and Painful Sensations (MAPPS) is an outline of a human body overlaid by a grid of 786 sensation pixels that was developed using the Qualtrics online survey platform, which can be recreated on any device capable of supporting a web-browser. Mouse clicks allow respondents to identify locations (i.e., grid pixels) on the manikin where they feel both pleasant and unpleasant sensations. Clicking once in any grid pixel turns that location blue, indicating a pleasant sensation. Clicking twice in any grid pixel turns that location red, indicating an unpleasant sensation. A ratio of pleasant to unpleasant sensations is derived from MAPPS.
Longer-Term Change in Pleasant Sensation Ratios | At baseline and posttreatment, approximately 1.5 months
  The Multidimensional Assessment of Pleasant and Painful Sensations (MAPPS) is an outline of a human body overlaid by a grid of 786 sensation pixels that was developed using the Qualtrics online survey platform, which can be recreated on any device capable of supporting a web-browser. Mouse clicks allow respondents to identify locations (i.e., grid pixels) on the manikin where they feel both pleasant and unpleasant sensations. Clicking once in any grid pixel turns that location blue, indicating a pleasant sensation. Clicking twice in any grid pixel turns that location red, indicating an unpleasant sensation. A ratio of pleasant to unpleasant sensations is derived from MAPPS.

SECONDARY OUTCOMES:
Change in Opioid Medication Desire | Immediately before and immediately after the final mindfulness training session, approximately 30 minutes
  Single-item Numeric Rating Scale (0-10), with 0 indicating no desire for opioid medication and 10 representing the an intense desire for opioid medication.
Change in Pain Intensity | Immediately before and immediately after the final mindfulness training session, approximately 30 minutes
  Single-item Numeric Rating Scale (0-10), with 0 indicating no pain and 10 representing the an most intense pain imaginable.
Change in Opioid Use | At baseline and 1-month follow-up, approximately 3 months
  Opioid Use will be assessed with a timeline follow-back procedure.
Change in Pain Functional Interference | At pretreatment and 1-month follow-up, approximately 3 months
  Pain functional interference will be assessed with the Brief Pain Inventory.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No